CLINICAL TRIAL: NCT02431312
Title: Phase I, Randomized, Open-Label, Active-Controlled, Dose Escalation Study to Evaluate the Safety, Tolerability & Immunogenicity of INO-1800 Alone or in Combination With INO-9112 Delivered IM Followed by EP in Select Nucleos(t)Ide Analogue-Treated, Chronic Hepatitis B Patients
Brief Title: Phase I Study of INO-1800 With or Without INO-9112 + EP in Chronic Hepatitis B Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HBV-001
Record Dates: First submitted 2015-04-21; First posted 2015-05-01 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Hepatitis B
Keywords: Chronic HBV; immunotherapy; DNA vaccine; electroporation
MeSH Terms: conditions — Hepatitis B | interventions — rocakinogene sifuplasmid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group A: low dose, standard regimen (Experimental): Participants received 3 or 4 doses of 0.3 mg INO-1800 delivered by EP in a standard regimen while continuing treatment with nucleos(t)ide analogue treatment.
  Interventions: Biological: INO-1800; Drug: Nucleos(t)ide Analogue Treatment
- Group A: mid dose, standard regimen (Experimental): Participants received 3 or 4 doses of 2 mg INO-1800 delivered by EP in a standard regimen while continuing treatment with nucleos(t)ide analogue treatment.
  Interventions: Biological: INO-1800; Drug: Nucleos(t)ide Analogue Treatment
- Group A: high dose, standard regimen (Experimental): Participants received 3 or 4 doses of 9 mg INO-1800 delivered by EP in a standard regimen while continuing treatment with nucleos(t)ide analogue treatment.
  Interventions: Biological: INO-1800; Drug: Nucleos(t)ide Analogue Treatment
- Group B: mid dose, standard regimen (Experimental): Participants received 3 or 4 doses of 2 mg INO-1800 + 0.25 mg INO-9112 delivered by EP in a standard regimen while continuing treatment with nucleos(t)ide analogue treatment.
  Interventions: Biological: INO-1800; Biological: INO-9112; Drug: Nucleos(t)ide Analogue Treatment
- Group B: high dose, standard regimen (Experimental): Participants received 3 or 4 doses of 9 mg INO-1800 + 0.25 mg INO-9112 delivered by EP in a standard regimen while continuing treatment with nucleos(t)ide analogue treatment.
  Interventions: Biological: INO-1800; Biological: INO-9112; Drug: Nucleos(t)ide Analogue Treatment
- Active Control: nucleos(t)ide analogue treatment (Active Comparator): Participants continued treatment with nucleos(t)ide analogue treatment.
  Interventions: Drug: Nucleos(t)ide Analogue Treatment

INTERVENTIONS:
Biological: INO-1800 — INO-1800 delivered by EP
  Arms: Group A: high dose, standard regimen; Group A: low dose, standard regimen; Group A: mid dose, standard regimen; Group B: high dose, standard regimen; Group B: mid dose, standard regimen
Biological: INO-9112 — INO-9112 delivered by EP
  Arms: Group B: high dose, standard regimen; Group B: mid dose, standard regimen
Drug: Nucleos(t)ide Analogue Treatment — Continued treatment with nucleos(t)ide analogue

SUMMARY:
This was an open-label study that evaluated the safety, tolerability, and immunogenicity of dose combinations of INO-1800 (DNA plasmids encoding Hepatitis B surface antigen [HBsAg] and Hepatitis B core antigen [HBcAg]) and INO-9112 (DNA plasmid encoding human interleukin 12) delivered by electroporation (EP) in 90 (ninety) nucleos(t)ide analogue treated participants.

ELIGIBILITY:
INCLUSION CRITERIA:

* Chronic Hepatitis B virus infection
* Negative for Hepatitis A IgM, C, D and HIV
* Liver biopsy, Fibroscan® or equivalent elastography-based test obtained within the past 6 months demonstrating liver disease without evidence of bridging fibrosis or cirrhosis supported by platelet count greater than the central laboratory LLN at screening
* Positive for Hepatitis B surface antigen (≥250 IU/mL at screening)
* Nucleos(t)ide treatment for at least 1 year with ongoing nucleos(t)ide analogue treatment at randomization
* HBV DNA <90 IU/mL for ≥6 months prior to randomization
* Screening laboratory values within normal range
* ALT ≤1.5x upper limit of normal (ULN) from 2 measurements separated by at least 14 days during the 6 months prior to randomization and ALT at screening ≤1.5x ULN
* AST, TBili, DBili, GGT, Alk Phos and albumin within normal range or judged to be not clinically significant by PI and medical monitor at screening
* For men and women who are not postmenopausal [i.e. ≥ 12 months of non-therapy-induced amenorrhea, confirmed by follicle stimulating hormone (FSH), if not on hormone replacement] or surgically sterile (vasectomy in males or absence of ovaries and/or uterus in females) agreement to remain abstinent or use 1 highly effective or combined contraceptive methods that result in a failure rate of < 1% per year during the treatment period and at least through week 12 after last dose

EXCLUSION CRITERIA:

* Pregnant or breastfeeding females
* Positive serum pregnancy test at screening or positive urine pregnancy test at randomization
* Use of topical corticosteroids at or near the intended administration site
* Autoimmune disorders, transplant recipients, other immunosuppression including any concurrent condition requiring the use of immunosuppressive/immunomodulating agents (eye drop-containing and infrequent inhaled corticosteroids are permissible)
* Need for systemic antiviral treatment (other than for chronic hepatitis B infection)
* Documented history or other evidence of decompensated liver disease (e.g., ascites, bleeding from esophageal varices, Child-Pugh clinical classification B or C)
* History of liver cirrhosis demonstrated by biopsy, Fibroscan® or equivalent elastography-based test
* History of other evidence of a medical condition associated with chronic liver disease [e.g., hemochromatosis, autoimmune hepatitis, alcoholic liver disease, non-alcoholic steatohepatitis (NASH), toxin exposure, thalassemia, etc.]
* Documented history or other evidence of metabolic liver disease within 1yr of randomization
* Abnormal renal function including serum creatinine >ULN or calculated creatinine clearance <70 mL/min (using the Cockcroft Gault formula)
* History of or suspicion of HCC
* Screening alpha fetoprotein ≥13 ng/mL
* Prior history or current malignancy other than adequately treated BCC, unless history of BCC is near intended administration site
* History of significant medical conditions [e.g., cardiac (including ventricular or supraventricular arrhythmias), renal disease, pulmonary, gastrointestinal, neurological]
* Significant acute infection (e.g., influenza, local infection) or any other clinically significant illness within 2 weeks of randomization
* Administration of any blood product within 3 mon of randomization
* History of seizures (unless seizure free for 5yrs)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
Safety Assessment (Composite of multiple measures: pain (VAS), adverse events, lab abnormalities, changes in vital signs) | Signing of ICF through up to 76 weeks following the first dose
  Composite outcome measure consisting of multiple measures, including:
  1. Local pain immediately after Study Treatment/EP and at select times using a visual analog scale (VAS) from 0 to 10, with 0 representing "No Pain" and 10 representing "Worst Pain"
  2. Frequency and severity of local and systemic events for at least 7 days after Study Treatment/EP
  3. Frequency and severity of laboratory abnormalities
  4. Frequency and severity of all adverse events
  5. Changes in vital signs

SECONDARY OUTCOMES:
Immunogenicity Assessment | Baseline (screening and first dose) and select points up to 76 weeks after the first dose
  Composite outcome measure consisting of multiple measures, including
  1. Breadth and Magnitude of antigen specific cellular immune responses
     * Interferon-ɣ ELISpot
     * Flow Cytometry for T-cell activation, cytolytic phenotype, memory phenotype
  2. Breadth and Magnitude of antigen specific ELISA
Viral/Antiviral Assessment | Screening and/or first dose and select points up to 76 weeks after the first dose
  Composite outcome measure consisting of multiple measures, including:
  1. Evaluate effect on HBsAg kinetics as measured in the quantitative HBsAg assay
  2. Evaluate effect on maintenance of HBV DNA suppression (< 90 IU/ml) as measured in the quantitative viral load assay

OTHER OUTCOMES:
Exploratory Assessment | Screening and/or first dose and select points up to 76 weeks after the first dose
  Composite outcome measure consisting of multiple measures, including:
  1. Relationship between immunogenicity and antiviral response
  2. Expression of individual markers potentially predictive of immunogenic and antiviral responses

CONTACTS AND LOCATIONS:
Overall Officials: ShuPing Yang, MD, PhD, Study Director — Inovio Pharmaceuticals
Locations (22):
- United States (7):
  - Research and Education, Inc., San Diego, California
  - University of Miami Schiff Center for Liver Disease, Miami, Florida
  - Northwell Health, Manhasset, New York
  - Mount Sinai - PRIME, New York, New York
  - UC Physicians Company, LLC/Division of Digestive Diseases, Cincinnati, Ohio
  - Philadelphia VA Medical Center, Philadelphia, Pennsylvania
  - Harbourview Medical Center, Seattle, Washington
- Australia (3):
  - Nepean Hospital, Kingswood, New South Wales
  - Mater Adult Hospital, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
- The University of Hong Kong, Hong Kong, Hong Kong
- Auckland City Hospital, Auckland, New Zealand
- The Medical City, Pasig, Philippines
- Singapore General Hospital, Singapore, Singapore
- Taiwan (5):
  - Chang Gung Memorial Hospital, Linkou District, Taoyuan County
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (3):
  - Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Tha Muang, Chiang Mai
  - Srinagarind Hospital, Khon Kaen, Muang District